CLINICAL TRIAL: NCT00161434
Title: A Randomized, Double-Blind, Placebo Controlled Crossover Trial Using Valacyclovir to Suppress HSV and HIV Shedding in HIV-1, HSV-2 Coinfected Persons
Brief Title: A Study of Valacyclovir to Suppress HSV and HIV Shedding in Coinfected Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Anna Wald, MD, MPH, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 02-6505-A; P01AI030731 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: HIV-1
MeSH Terms: conditions — Herpes Simplex; HIV Infections | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: valacyclovir
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: valacyclovir — 1 gram daily for 8 weeks
  Other Names: Valtrex
  Arms: 1
Drug: placebo — matching placebo for 8 weeks
  Arms: 2

SUMMARY:
The primary objective of this research study is to assess if daily valacyclovir therapy for suppression of HSV-2 reactivation is associated with a decrease in mucosal HIV shedding in individuals co-infected with both HSV-2 and HIV.

DETAILED DESCRIPTION:
Sexually transmitted diseases and genital ulcer disease (GUD) contribute significantly to the spread of HIV, as their presence is associated with higher rates of HIV acquisition in susceptible individuals. Herpes simplex virus-2 (HSV-2) is a major cause of GUD in developed and developing countries.

The primary objective of this research study is to assess if daily valacyclovir therapy for suppression of HSV-2 reactivation is associated with a decrease in mucosal HIV shedding in individuals co-infected with both HSV-2 and HIV.

This study is a randomized, double-blind, placebo-controlled, crossover trial. Sixty men who have sex with men (MSM) will be randomized to first receive either valacyclovir, 1 gram once a day, or matching placebo for 8 weeks. After a 2-week washout period during which all participants receive placebo, subjects then switch to the other treatment for the next 8 weeks.

At screening, informed consent is obtained and individuals will have blood drawn to test antibody status to HIV and HSV and well as to monitor CD4 count and plasma HIV RNA determination. At enrollment, oral, genital, and rectal specimens are obtained and additional blood is drawn. Participants are given a two-week supply of study medication and are instructed on the technique of collecting daily home samples and completing a diary. Following enrollment, they are asked to collect daily home oral and genital samples, as well as semen samples twice a week, for the full 18 weeks of the study. Participants return to the clinic three times per week for follow-up, for collection of oral and rectal specimens, and additional study medication. Rectal Biopsy is performed at weeks 8 and 18 for those individuals that signed the additional rectal biopsy consent form.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive and HSV-2 seropositive
* MSM (men having sex with men)
* 18 years old or older

Exclusion Criteria:

* Known history of adverse reaction to acyclovir or valacyclovir
* Planned open label use of acyclovir, valacyclovir or famciclovir

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess reduction in mucosal HIV shedding associated with daily valacyclovir for suppression of HSV-2 reactivation. | 18 weeks

SECONDARY OUTCOMES:
To quantify increase in rectal and pharyngeal HIV-1 shedding associated with HSV-1 and HSV-2 reactivation. To determine reduction in systemic HIV RNA during valacyclovir therapy. To evaluate reduction in inflammatory cells and HIV replication. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Virology Research Clinic, Seattle, Washington, United States